CLINICAL TRIAL: NCT04831034
Title: 68Ga-DOTA/NOTA-FAPI PET/CT in Patients With Various Fibrotic Disease
Brief Title: 68Ga-FAPI PET/CT in Patients With Various Fibrotic Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian7
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Fibrosis; Positron-Emission Tomography
MeSH Terms: conditions — Fibrosis | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-04 (Experimental): Each subject receive a single intravenous injection of 68Ga-DOTA/NOTA-FAPI-04, and undergo PET/CT imaging within the specificed time.
  Interventions: Drug: 68Ga-FAPI-04

INTERVENTIONS:
Drug: 68Ga-FAPI-04 — Each subject receive a single intravenous injection of 68Ga-FAPI-04, and undergo PET/CT scanning within the specified time.

SUMMARY:
To evaluate the potential value of 68Ga-FAPI-04 positron emission tomography/ computed tomography (PET/CT) for the diagnosis and prognosis in fibrotic disease

DETAILED DESCRIPTION:
Subjects with fibrotic disease underwent 68Ga-FAPI-04 PET/CT scanning. Fibrosis lesion uptake was quantified by the maximum standard uptake value (SUVmax). Subjects also received the conventional clinical assessment for liver fibrosis, such as magnetic resonance imaging(MRI) , biopsy and blood biochemical indexes (BBI) testing. The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga-FAPI-04 PET/CT, MRI and BBI were calculated and compared to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or order)
* patients with suspected or new diagnosed fibrotic disease (supporting evidence may include , BBI, MRI, CT and pathology report)
* patients who had scheduled 68Ga-FAPI-04 PET/CT scan
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee

Exclusion Criteria:

* patients with pregnancy
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 68Ga-DOTA/NOTA-FAPI-04 for each target lesion of subject.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of 68Ga-DOTA/NOTA-FAPI-04 PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No